CLINICAL TRIAL: NCT07171333
Title: Role of Computer-Aided Detection Colonoscopy in Polyp Detection Rate: an Italian Multi-Center Randomized Study (CADEC)
Brief Title: Role of Computer-Aided Detection Colonoscopy in Polyp Detection Rate
Acronym: CADEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gian Eugenio Tontini (Other)
Collaborators: Pentax Medical (Industry)
Responsible Party: Sponsor-Investigator, Gian Eugenio Tontini, Prof., Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Organization: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OSMAMI-15/09/2022-0042892-U
Record Dates: First submitted 2025-08-30; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Polyps
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- CADe+ (Experimental): colonoscopy with CADe system
  Interventions: Device: Colonoscopy with CADe system
- CADe- (No Intervention): colonoscopy without CADe system

INTERVENTIONS:
Device: Colonoscopy with CADe system — Patients in the CADe+ arm underwent colonoscopy with CADe DISCOVERY™ (PENTAX Medical, Tokyo, Japan), an AI-driven tool highlighting suspected lesions in real-time, through a light-blue box. The final lesion characterization remained the endoscopist's responsibility.
  Arms: CADe+

SUMMARY:
High-definition (HD) colonoscopy is the gold standard for early diagnosis and treatment of lower gastrointestinal neoplasms, with the adenoma detection rate (ADR) serving as a key quality indicator due to its inverse correlation with colorectal cancer incidence. ADR is influenced by operator expertise, fatigue, and human error, which may be mitigated by advanced imaging technologies such as computer-aided detection (CADe). CADe systems provide real-time visual and auditory alerts for suspected polyps and have been shown to increase ADR, though their effectiveness under different operator conditions (high- vs. low-volume, fatigue-related performance, impact on polyp detection rate [PDR] and withdrawal time) remains unclear. This multicenter, prospective, national, open-label randomized trial (6 Italian centers) will compare HD-Iscan colonoscopy with and without CADe assistance (1:1 allocation), with primary endpoint ADR and secondary endpoints including PDR, withdrawal time, and performance stratified by operator fatigue. Eligible patients (aged 40-80, undergoing screening, surveillance, or diagnostic colonoscopy) will be recruited consecutively, with exclusions for prior colonic resection, recent diverticulitis, inflammatory bowel disease, familial polyposis, inadequate bowel preparation, complete colonoscopy within 5 years, inability to consent, or unsafe ongoing antithrombotic therapy. Colonoscopies will follow ESGE guidelines with standard split-dose PEG preparation; all polyps will be resected and documented. Operator allocation to high- (≥200 colonoscopies/year) or low-volume (<200/year) groups will follow routine clinical scheduling, with stratified analyses performed. The trial involves no investigational drugs or additional invasive procedures, and no adverse events are anticipated beyond those inherent to colonoscopy.

ELIGIBILITY:
Inclusion criteria:

* Age 40-80 years, any sex
* Indication for screening, surveillance, or diagnostic colonoscopy (e.g., anemia, abdominal symptoms)
* Written informed consent

Exclusion criteria:

* Previous (even partial) colon resection or colonic stenosis
* Acute diverticulitis within 4 weeks
* Inflammatory bowel disease, familial adenomatous polyposis, or microscopic colitis
* Complete colonoscopy within 5 years
* Inadequate suspension of antithrombotic/antiplatelet therapy (per ESGE guidelines)
* Inability to provide consent
* Inadequate bowel preparation (Boston Bowel Preparation Scale <2 in any segment)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate | 2 weeks
  Adenoma detection rate (ADR) is the percentage of patients with at least one histologically proven adenoma or carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Gian Eugenio Tontini, MD, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Access Criteria: Researchers who provide a methodologically sound proposal.